CLINICAL TRIAL: NCT03858660
Title: Physical Examination for Health Management in Elderly
Brief Title: Clinical Applications of a Smart Physical Examination System for the Health Management in Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807156DINC
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Conditions Influencing Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Healthy elderly No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aging usually results in a decline in motor function. However, the elderly tend to refuse the regular health examination because of travel issues or lack of self-health awareness. Examination unit also has difficulty to intensively track and instant feedback on the health status of the elderly due to insufficient manpower. If the elderly go to the hospital only when the health problem is getting worse, his/her health is often irreversible and the cost of medical care would be increased. It is therefore an essential issue for the early detection of functional changes in the elderly to prevent the deterioration of the health and function. Currently, the telemedicine cares provided by hospitals are not universal due to the out-of-date legislation and non-successful business model. The wearing and operation issues of the wearable devices used for health management are still a gap affecting the acceptance of the elderly. Accordingly, the objective of this project is to develop a handy and easy-to-use smart physical examination system for the elderly. With the use of motion-sensing and big data analysis technology, the non-contact professional and intelligent assessment could simplify the general health checkup procedures to promote the health management and to reduce the manpower cost of health care. The ultimate goal is to realize a commercial product aiming at the silver hair market with functional advantages to meet the unmet needs of health management in the elderly.

DETAILED DESCRIPTION:
[Introduction] Aging usually results in a decline of motor function. However, elderly tends to refuse the regular health examination because of travel issues or lack of self-health awareness. Examination unit also has difficulty to intensively track and instantly feedback the health status of elderly due to insufficient manpower. If elderly goes to the hospital only when the health problem is getting worse, his/her health is often irreversible and the cost of medical care would be increased. It is therefore an essential issue for the early detection of functional changes in elderly to prevent the deterioration of the health and function. Currently, the telemedicine cares provided by hospitals are not universal due to the out-of-date legislation and non-successful business model. The wearing and operation issues of the wearable devices used for health management are still a gap affecting the acceptance of elderly. Accordingly, the objective of this project is to develop a handy and easy-to-use smart physical examination system targeted on the unmet need of the elderly. With the use of motion-sensing and big data analysis technology, the non-contact professional and intelligent assessment could simplify the general health checkup procedures to promote the health management and to reduce the manpower cost of health care. The ultimate goal is to realize a commercial product aiming at the silver hair market with functional advantages to meet the unmet needs of health management in elderly.

In this study, a new type of home-based health assessment platform will be proposed. The main purpose is to help the elderly who may not be able to go to the hospital or health unit for regular health check because of inconvenience to physical activity. The current health assessment mode is also insufficient because Human and resource could not provide a more intensive frequency of health testing. The physical condition of the elderly may rapidly decline into a systemic disability due to some minor diseases. Therefore, the current limited resource inspection mode cannot effectively monitor and recover the elderly's physical condition. The home-based health assessment platform developed in this study can evaluate the user's health status in hospitals, communities, or home environments. The non-contact evaluation method allows users to start testing without wearing any device, which can effectively improve The user's acceptance of health testing and rapid grading of the user's health will also help to further design a personalized rehabilitation training program in the future.

[Method]

Subject:

Inclusion criteria: 1) aged between 55-85 years old. 2) normal upper extremity function. 3) walk for at least 10 meters without help.

Exclusion criteria: 1) any disease that could affect balance. 2) deficits in vision or hearing. 3) mental issues preclude from the understanding of the protocol.

Protocol:

1. Basic information: including gender, age, height, leg length, weight, medical history, medication, etc.
2. Clinical functional assessment: The results of following tests evaluated by the Kinect-based health management platform will be compared with those of the physical examination conducted by experts such as clinicians and therapists.

   i. Flexibility test: The subjects sit in a chair with no backrest and backrest. One foot bent stably on the ground and one foot extended forward (knee joint must be straight). The heel hits the ground and the foot was in neutral position. They are then asked to overlap the hands and straighten the upper body forward slowly, trying to touch the toes in the middle pointing and holding for 2 seconds. The distance between the middle finger and the toes is then measured. The test are repeated twice and the better measured value will be recorded.

   ii. Endurance test: evaluated by the 2-minute stepping test. iii. Muscle strength: Upper limb strength is assessed using a 30-second arm curl test. And the lower limb strength is assessed by the 30-second sit-to-stand test.

   iv. Balance test: The subjects are asked to stand on the force plate looking straight ahead with feet in shoulder width. There are two kinds of standing test situations: i) single leg standing for a maximum of 60 seconds; ii) forward reaching as the arms straight and parallel to the ground and remain in the maximum extended position for two seconds.

   v. Questionnaire: EuroQOL-5D will be used to evaluate their quality of life.
3. Data analysis: The concurrent validity of the Kinect-based health management platform will be analyzed by the Pearson Correlation. And the balance parameters will be evaluated by the movement of center of the pressure.
4. Adverse reactions and management: All the tests are non-invasive, so we won't expect any major side effects. If the patient feels uncomfortable or feels dizzy during the fitness test, he can stop the test, lie down and rest at any time, and the on-site medical staff will monitor their breathing, heartbeat, and blood pressure to assess whether additional treatment is required.

ELIGIBILITY:
Inclusion Criteria:

* Normal upper extremity function
* Walk for at least 10 meters without help

Exclusion Criteria:

* Any conditions that could affect the balance function
* Deficits in vision or hearing
* Mental conditions that preclude the understanding of the protocol

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-09-18 (Estimated); Study Completion 2019-09-18 (Estimated)

PRIMARY OUTCOMES:
Balance performance | 2 minutes
  Forward reaching test
Fitness | 2 minutes
  flexibility test
Lower extremity function | 2 minutes
  2 minute step
Muscle force | 2 minutes
  weight lifting
Endurence | 2 minutes
  30sec sit-to-stand
Questionaire | 5 minutes
  EuroQOL-5D

CONTACTS AND LOCATIONS:
Overall Officials: Der-Sheng Han, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No